CLINICAL TRIAL: NCT03270826
Title: Physiological Behavior of Respiratory Maneuvers Through Electrical Impedance Tomography and Optoelectronic Plethymography
Brief Title: Physiological Behavior of Respiratory Maneuvers
Status: Completed | Type: Observational
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Cláudia Thais Pereira Pinto, Principal Investigator, Universidade Federal de Pernambuco
Other Study IDs: 23031990
Record Dates: First submitted 2017-06-16; First posted 2017-09-01 (Actual); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Introduction: new methods of evaluation of respiratory function, such as electrical impedance tomography (EIT) and optoelectronic plethysmography (OEP), have been used to measure regional pulmonary ventilation and the variation of tricompartmental volumes of the thoracic cavity, respectively. Analysis of these instruments during maximal respiratory maneuvers with monitoring of esophageal pressure may probably provide additional information on the physiological behavior of the cardiorespiratory system during EIT and OEP maneuvers. Objectives: To describe the physiological behavior of maximal respiratory maneuvers through the electrical impedance tomography and optoelectronic plethysmography in healthy men.

METHODS: This is a cross-sectional study involving 10 healthy male volunteers. The development of the method will take place in 3 stages. The first step corresponds to the characterization of the inspiratory and expiratory curves in the respiratory cycle generated by the impedance variation (ΔZ), the mobility of the chest wall and the pulmonary volume curve during maximal respiratory maneuvers. 2nd stage: verification of the correlation between the variables Step 3: Estimate the dislocated blood volume of the lung through previous analyzes.

DETAILED DESCRIPTION:
The physiological repercussions resulting from the maximal respiratory maneuvers together with the synchronized analysis of the chest cavity mobility, pulmonary volume , pulmonary impedance and measurement of Oesophageal pressure is not known. Therefore, this study aims to describe the physiological behavior of maximal respiratory maneuvers through the synchronization between electrical impedance tomography and optoelectronic plethysmography in healthy men.

ELIGIBILITY:
Inclusion Criteria:

* Will be included in the study male volunteers,
* BMI greater than or equal to 18.5 and less than 25 kg / m2, considered adequate or eutrophic (MS, 2011)
* Chest circumference between 44 and 55 cm if fitted to the electrical impedance tomography (EIT) strap size P or M;
* systolic blood pressure lower than 140 mmHg and greater than 100 mmHg
* diastolic blood pressure greater than 60 mmHg and lower than 90 mmHg (VI Brazilian Guidelines for Hypertension, 2010)
* without reports of cardiovascular or pulmonary diseases and symptoms Last month.

Exclusion Criteria:

* Volunteers who refuse to participate in the study will be excluded from the survey;
* Presence of cardiac dysfunction assessed by echocardiography;
* Altered pulmonary function by spirometry (PEREIRA et al, 2001) and manovacuometry according to predicted values for healthy individuals (PESSOA et al, 2014).
* Presence of tissue injury in the thorax;
* Dysautonomia that may indicate dysfunction of the autonomic nervous system (ANS), with following clinical manifestations: seizures; epilepsy; Anhydrosis and hyperhidrosis; Neurogenic bladder (CASTRO et al, 1992); (Stewart et al., 2004 and 2005)
* individuals who donated blood or had significant blood loss within 30 days prior to the start of the study (Navarro et al, 1997).

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study sample will be composed of healthy male volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2017-04-07 (Actual); Primary Completion 2018-02-20 (Actual); Study Completion 2018-03-23 (Actual)

PRIMARY OUTCOMES:
Displacement of blood volume of the lung | 09/03/2018
  Volume displacement per unit time measured by electrical impedance tomography through the impedance variation in Ohm (Ω).

SECONDARY OUTCOMES:
Variation of pulmonary electrical impedance | 09/03/2018
  Variation between the final and initial impedance measured by electrical impedance tomography through the impedance variation in Ohm (Ω).

OTHER OUTCOMES:
Lung volume | 09/03/2018
  Measurement of the amount of air that the lungs may contain at various points in the respiratory cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Cláudia Thais Pinto, Ms, Principal Investigator — UFPE
Locations (1):
- Universidade Federal de Pernambuco, Recife, PE - Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: No